CLINICAL TRIAL: NCT00823745
Title: A Phase 1 Study To Evaluate The Metabolism And Excretion Of [14C] PF-00868554 In Healthy Adult Male Subjects
Brief Title: Radiolabel ADME (Absorption, Distribution, Metabolism, and Excretion) Study Of [14C] PF-00868554 In Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A8121013
Record Dates: First submitted 2009-01-07; First posted 2009-01-16 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: HCV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): [14C]-PF-00868554
  Interventions: Drug: [14C]-PF-00868554

INTERVENTIONS:
Drug: [14C]-PF-00868554 — solution, single dose

SUMMARY:
This is a phase 1 study to assess the routes of elimination of a single oral dose of [14C] PF-00868554 and to characterize the metabolic profile following single dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Male, healthy volunteers.

Exclusion Criteria:

* Females.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The amount of radioactivity recovered in urine and feces, as a percent of the dose. | 7 weeks
The amount of PF-00868554, expressed as a percent of total radioactivity, in plasma, urine, and feces. | 7 weeks
Identification and determination of relative abundance of the metabolites of PF-00868554 in plasma, urine, and feces. | 7 weeks
PK parameters: AUClast, AUCinf, maximum concentration (Cmax), time of maximum concentration (Tmax), and half-life (t1/2) to describe the single dose PK of a) total radioactivity in blood; b) total radioactivity in plasma; c) PF-00868554 in plasma. | 7 weeks

SECONDARY OUTCOMES:
Safety endpoints including adverse events, clinical laboratory tests, vital signs and ECGs. | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Tacoma, Washington, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8121013&StudyName=Radiolabel%20ADME%20%28Absorption%2C%20Distribution%2C%20Metabolism%2C%20and%20Excretion%29%20Study%20Of%20%5B14C%5D%20PF-00868554%20In%20Healthy%20Adult%20Male%20Subjects